CLINICAL TRIAL: NCT00396760
Title: The Influence of High-Dose Aprotinin and Tranexamic Acid on Bleeding Tendency and Allogeneic Blood Transfusion in Patients Undergoing Primary Aortic Valve Replacement or Coronary Artery Revascularization
Brief Title: Comparison of Aprotinin and Tranexamic Acid in Routine Cardiac Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: German Heart Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1172/04
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2006-11

CONDITIONS: Bleeding and Cardiac Surgery; Allogeneic Blood Transfusion; Aortic Valve Replacement; Coronary Artery Bypass Graft Surgery
Keywords: cardiac surgery; blood transfusion; antifibrinolytics; aprotinin; tranexamic acid
MeSH Terms: conditions — Hemorrhage | interventions — Aprotinin; Tranexamic Acid

INTERVENTIONS:
Drug: aprotinin or tranexamic acid

SUMMARY:
The hypothesis of this study is that the antifibrinolytic drugs aprotinin and tranexamic acid equally influence bleeding tendency and transfusion requirement in patients undergoing first time cardiac procedures with a low risk of increased postoperative bleeding.Only patients undergoing first time CABG or first time aortic valve replacement are included in this study.

DETAILED DESCRIPTION:
Excessive bleeding during and after cardiac surgery is a serious complication. It exposes patients to the risk of allogeneic blood transfusion or other blood products and the risk of mediastinal re-exploration.Antifibrinolytic drugs like aprotinin and tranexamic acid are proven to reduce bleeding tendency and transfusion requirement in cardiac surgery. The efficacy of these drugs is proven, especially for the unspecific proteinase inhibitor aprotinin, however, there are concerns about the safety and the high costs of this drug. There are only limited head-to-head comparisons of these two drugs.

In this double-blind, prospective, controlled study the efficacy of aprotinin and tranexamic acid is compared. Primary outcome is the 24 hours postoperative drainage blood loss and the percentage of patients requiring allogeneic blood transfusion during the hospital stay. Subgroups of patients undergoing CABG surgery or aortic valve replacement are predefined for combined and separate data analysis.The power of the study is calculated for this subgroup-analysis.

Secondary outcome measurements are molecular marker of activation of hemostasis up to the 5th postoperative day.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* Patients undergoing primary CABG or Aortic valve replacement surgery

Exclusion Criteria:

* Previous sternotomy
* OPCAB surgery
* urgent/emergency operation
* Coumadin treatment
* previous aprotinin exposure
* preoperative renal impairment (Creatinine > 2 mg/dL)
* patients refusing blood transfusions
* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2005-01; Study Completion 2006-07

PRIMARY OUTCOMES:
24 hours postoperative drainage blood loss
incidence of allogeneic blood transfusion

SECONDARY OUTCOMES:
activation of fibrinolysis and hemostasis
impairment of renal function

CONTACTS AND LOCATIONS:
Overall Officials: Wulf Dietrich, MD, PhD, Principal Investigator — Department of Anesthesiology, German Heart Center Munich
Locations (1):
- German Heart Center Munich, Munich, Munich, Germany

REFERENCES:
- [Background] Diprose P, Herbertson MJ, O'Shaughnessy D, Deakin CD, Gill RS. Reducing allogeneic transfusion in cardiac surgery: a randomized double-blind placebo-controlled trial of antifibrinolytic therapies used in addition to intra-operative cell salvage. Br J Anaesth. 2005 Mar;94(3):271-8. doi: 10.1093/bja/aei044. Epub 2004 Dec 10. PMID 15591329
- [Background] Henry DA, Moxey AJ, Carless PA, O'Connell D, McClelland B, Henderson KM, Sly K, Laupacis A, Fergusson D. Anti-fibrinolytic use for minimising perioperative allogeneic blood transfusion. Cochrane Database Syst Rev. 2001;(1):CD001886. doi: 10.1002/14651858.CD001886. PMID 11279735
- [Background] Royston D, Levy JH, Fitch J, Dietrich W, Body SC, Murkin JM, Spiess BD, Nadel A. Full-dose aprotinin use in coronary artery bypass graft surgery: an analysis of perioperative pharmacotherapy and patient outcomes. Anesth Analg. 2006 Nov;103(5):1082-8. doi: 10.1213/01.ane.0000238447.74029.f5. PMID 17056936
- [Background] Dietrich W, Busley R, Kriner M. High-dose aprotinin in cardiac surgery: is high-dose high enough? An analysis of 8281 cardiac surgical patients treated with aprotinin. Anesth Analg. 2006 Nov;103(5):1074-81. doi: 10.1213/01.ane.0000238446.30034.c8. PMID 17056935
- [Derived] Lison S, Dietrich W, Braun S, Boehm J, Schuster T, Englhard A, Perchuc A, Spannagl M, Busley R. Enhanced thrombin generation after cardiopulmonary bypass surgery. Anesth Analg. 2011 Jan;112(1):37-45. doi: 10.1213/ANE.0b013e3181fc6df0. Epub 2010 Dec 2. PMID 21127274
- [Derived] Dietrich W, Spannagl M, Boehm J, Hauner K, Braun S, Schuster T, Busley R. Tranexamic acid and aprotinin in primary cardiac operations: an analysis of 220 cardiac surgical patients treated with tranexamic acid or aprotinin. Anesth Analg. 2008 Nov;107(5):1469-78. doi: 10.1213/ane.0b013e318182252b. PMID 18931201